CLINICAL TRIAL: NCT04061798
Title: ACTION-1: ACT Guided Heparinization During Open Abdominal Aortic Aneurysm Repair, a Randomised Trial.
Brief Title: ACT Guided Heparinization During Open Abdominal Aortic Aneurysm Repair.
Acronym: ACTION-1
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Futility
Sponsor: Dijklander Ziekenhuis (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Amsterdam UMC, location VUmc (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Arno Wiersema, MD, PhD, Vascular Surgeon, Dijklander Ziekenhuis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL-66759
Record Dates: First submitted 2019-08-18; First posted 2019-08-20 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Abdominal Aortic Aneurysm; Surgery; Arterial Disease
Keywords: ACT guided heparinization in open aortic surgery
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Intervention Model Description: Intervention group:
  Heparin is given to reach an ACT of 200-220 seconds. At the start of the procedure, before any heparin is given, a baseline ACT measurement is performed. 3-5 minutes before clamping of the aorta 100 IU/kg bodyweight of heparin is administrated intravenously. 5 minutes after administration of heparin, ACT measurement is performed.
  Comparative group:
  A single dose of 5 000 IU of heparin is given 3-5 minutes before clamping of the aorta. No ACT measurements are performed, except for one ACT measurement after re-establishing blood flow and removing all clamps.
Who Masked: Participant
Masking Description: Patients will be randomized using a computerized program (CASTOR EDC) with a random block size of a maximum of 8. The randomization will be stratified by participating centre. The participant is blinded to the allocated treatment.
  Separate evaluation of results and if complications can be labelled as TEC, will be performed by an Independent Central Adjudication Committee. The 3 members of this Committee will be blinded to the allocated treatment.
  Since the care provider and investigator have to do the ACT measuring, it is impossible to blind them to the allocated treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT guided heparinization (Experimental): Heparin is given to reach an ACT of 200-220 seconds. At the start of the procedure, before any heparin is given, a baseline ACT measurement is performed. 3-5 minutes before clamping of the aorta 100 IU/kg bodyweight of heparin is administrated intravenously. 5 minutes after administration of heparin, ACT measurement is performed.
  Interventions: Drug: ACT guided heparinization
- 5 000 IU of heparin (Active Comparator): A single dose of 5 000 IU of heparin is given 3-5 minutes before clamping of the aorta. No ACT measurements are performed, except for one ACT measurement after re-establishing blood flow and removing all clamps. Depending on that ACT value near the end of surgery, the local protamine can be given to neutralize the effect of heparin. Only on clarified indications extra doses of heparin or protamine are permitted, at the discretion of the attending vascular surgeon. Indications could be clot formation intravascular or in a prosthesis, excessive bleeding or prolonged operation duration. Deviations from protocol should be clearly stated with reasoning in the operative report.
  Interventions: Drug: 5 000 IU of heparin

INTERVENTIONS:
Drug: ACT guided heparinization — If the ACT is <180 sec., an additional dose of heparin of 60 IU/kg is administered. If the ACT is 180-200 sec., 30 IU/kg.
  If the ACT is >200 sec., no extra heparin is given. 5 min. after every administration of heparin the ACT is measured. If the ACT is >200 sec, the next ACT measurement is performed every 30 min., until the end of the procedure or until new heparin administration is required. After each new dose of heparin, an ACT measurement is performed after 5 min. and the above- described protocol of ACT measurements will be repeated. After re-establishing blood flow and removing all clamps, the ACT is measured.
  If the ACT at closure is 200-250 sec., 2500 IU of protamine should be administered. If >250 sec., 5000 IU protamine. If 180-200 sec., 1000 IU protamine. 5 min. after the administration of protamine, the ACT is measured. The ACT should preferably be below 180 sec. If the ACT is still more than 200 sec., protamine should be administered again.
  Arms: ACT guided heparinization
Drug: 5 000 IU of heparin — A single dose of 5 000 IU of heparin is given 3-5 min before clamping of the aorta. No ACT measurements are performed, except for one ACT measurement after re-establishing blood flow and removing all clamps. Only on clarified indications extra doses of heparin or protamine are permitted, at the discretion of the attending vascular surgeon. Indications could be clot formation intravascular or in a prosthesis, excessive bleeding or prolonged operation duration. Deviations from protocol should be clearly stated with reasoning in the operative report.
  If the ACT at closure is between 200 and 250 s, 2500 IU protamine should be administered. If the ACT is higher than 250 s, 5000 IU protamine should be administered. If the ACT is between 180 and 200 s, 1000 IU protamine should be administered. Five minutes after the administration of protamine, the ACT is measured. The ACT should preferably be below 180 s. If the ACT is still more than 200 s, protamine should be administered again.
  Arms: 5 000 IU of heparin

SUMMARY:
Aim of the ACTION-1 study is to determine whether ACT guided heparinization decreases thrombo-embolic complications (TEC) and mortality after elective open AAA surgery, without causing more bleeding complications.

DETAILED DESCRIPTION:
Heparin is used during open abdominal aortic aneurysm (AAA) surgery to reduce thrombo-embolic complications (TEC): such as myocardial infarction, stroke, peripheral embolic events and the related mortality. On the other hand, heparin may increase blood loss, causing harm for the patient.

Heparin has an unpredictable effect in the individual patient. The effect of heparin can be measured by using the Activated Clotting Time (ACT). ACT measurement in open AAA repair could be introduced to ensure the individual patient of safe, tailor-made anticoagulation with a goal ACT of 200-220 seconds. A randomized controlled trial (RCT) has to prove that ACT guided heparinization would result in fewer TEC and lower mortality than a standardized bolus of heparin of 5 000 international units (IU), the current gold standard. ACT guided heparinization results in higher doses of heparin during operation and this should not result in significantly more bleeding complications of importance.

The ACTION-1 study will evaluate the effect of weight dosed heparinization during open abdominal aortic aneurysm surgery.The study will be an international multi-centre single blind randomized controlled trial. Patients will be randomized using a computerized program (CASTOR EDC) with a random block size of a maximum of 8. The randomization will be stratified by participating centre. Separate evaluation of results and if complications can be labelled as TEC, will be performed by an Independent Central Adjudication Committee. The 3 members of this Committee will be blinded with regard to if the patient was randomized for ACT guided heparinization or standard bolus of 5 000 IU without ACT measurements.

In the intervention group, heparin is given to reach an ACT of 200-220 seconds. Based on the ACT, an additional dose of heparin will be administered. Five minutes after every administration of heparin the ACT is measured. If the ACT is 200 seconds or longer, the next ACT measurement is performed every 30 minutes, until the end of the procedure or until new heparin administration is required (because of ACT < 200 seconds). Depending on the ACT value near the end of surgery, protamine will be given to neutralize the effect of heparin.

In the comparative group, a single dose of 5 000 IU of heparin will be given 3-5 minutes before clamping of the aorta. No ACT measurements will be performed, except for one ACT measurement after re-establishing blood flow and removing all clamps. Depending on that ACT value near the end of surgery, the local protamine can be given to neutralize the effect of heparin.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak and read in local language of trial hospital.
* Patients older than 18 years scheduled for elective, open repair of an iliac or abdominal aortic aneurysm distal of the Superior Mesenteric Artery (SMA) (DSAA segment C).
* Implantation of a tube or bifurcation prosthesis.
* Trans-abdominal or retroperitoneal surgical approach of aneurysm.
* Able and willing to provide written informed consent.

Exclusion Criteria:

* Not able to provide written informed consent.
* Previous open or endovascular intervention on the abdominal aorta (previous surgery on other parts of the aorta or iliac arteries is not an exclusion criterion).
* History of coagulation disorders, heparin induced thrombocytopenia (HIT), allergy for heparin or thrombocyte pathology.
* Impaired renal function with EGFR below 30 ml/min.
* Acute open AAA surgery.
* Hybrid interventions.
* Connective tissue disorders.
* Dual anti-platelet therapy, which cannot be discontinued.
* Life expectancy less than 2 years.
* Inflammatory, mycotic or infected aneurysms.
* Allergy for protamine or fish protein

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2024-04-13 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Combined incidence of all thrombo-embolic complications (TEC) and all-cause mortality. | Within 30 days or during the same admission in hospital
  TEC are any complication as caused by thrombus or embolus perioperatively, including but not exclusively: myocardial infarction, leg ischemia, deep venous thrombosis, colon ischemia, transient ischemic attack (TIA)/stroke, graft thrombosis, peroperative thrombus requiring embolectomy or redo of an anastomosis, thrombus or embolus in organs or lower limbs and other peripheral thrombosis. Incidence of bleeding complications according to European multicenter study on Coronary Artery Bypass Grafting (E-CABG) classification, grade 1 and higher: per- or postoperative transfusion of 2 or more units of red blood cells, transfusion of platelets, transfusion of fresh frozen plasma or reoperation for bleeding during hospital stay.

SECONDARY OUTCOMES:
Complications (non-TEC). | Within 30 days or during the same admission in hospital
  All complications requiring re-operation, longer hospital stay, all other complications. Incidence of kidney injury as defined by RIFLE criteria: rise of serum creatinine > 100% or decrease of estimated Glomerular Filtration Rate (eGFR) with 50%.32 Allergic reactions. ACT values (in intervention group), total heparin administration, protamine administration. Peroperative blood loss, blood transfusions either autologous or homologous, other blood products administration, total operative time, aortic clamping time, use of adjunctive haemostatic products, length of hospital (including ICU) stay. Health status as measured with the EQ-5D-5L. Economic and healthcare costs evaluation by the institute for Medical Technology Assessment (iMTA) Medical Consumption Questionnaire(IMCQ) and iMTA Productivity Cost Questionnaire (IPCQ) and addition of out-of-pocket expenses.

CONTACTS AND LOCATIONS:
Locations (22):
- Germany (2):
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Krankenhaus Barmherzige Brüder, Regensburg
- Netherlands (20):
  - Treant Zorggroep, Emmen, Drenthe
  - Gelre Ziekenhuizen, Apeldoorn, Gelderland
  - Rijnstate, Arnhem, Gelderland
  - Slingeland Ziekenhuis, Doetinchem, Gelderland
  - Elisabeth TweeSteden Ziekenhuis, Tilburg, Noord-Braband
  - Amphia, Breda, North Brabant
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - AUMC Location VUmc, Amsterdam, North Holland
  - AUMC Location AMC, Amsterdam, North Holland
  - Dijklander Ziekenhuis, Hoorn, North Holland
  - Medisch Spectrum Twente, Enschede, Overijssel
  - Isala, Zwolle, Overijssel
  - Groene Hart, Gouda, South Holland
  - Leiden Universitair Medisch Centrum, Leiden, South Holland
  - Alrijne, Leiderdorp, South Holland
  - Maasstad Ziekenhuis, Rotterdam, South Holland
  - Haaglanden Medisch Centrum, The Hague, South Holland
  - Ziekenhuisgroep Twente, Almelo
  - Universitair Medisch Centrum Groningen, Groningen
  - St. Antonius ziekenhuis, Nieuwegein

IPD SHARING:
Plan to Share IPD: Yes
under pre-defined conditions and contract
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after data lock, 07-2024
Access Criteria: contract with pre-defined criteria according to government regulation concerning science research

REFERENCES:
- [Background] Burgers LT, Vahl AC, Severens JL, Wiersema AM, Cuypers PW, Verhagen HJ, Redekop WK. Cost-effectiveness of Elective Endovascular Aneurysm Repair Versus Open Surgical Repair of Abdominal Aortic Aneurysms. Eur J Vasc Endovasc Surg. 2016 Jul;52(1):29-40. doi: 10.1016/j.ejvs.2016.03.001. Epub 2016 Apr 23. PMID 27118618
- [Background] Behrendt CA, Sedrakyan A, Riess HC, Heidemann F, Kolbel T, Petersen J, Debus ES. Short-term and long-term results of endovascular and open repair of abdominal aortic aneurysms in Germany. J Vasc Surg. 2017 Dec;66(6):1704-1711.e3. doi: 10.1016/j.jvs.2017.04.040. Epub 2017 Aug 7. PMID 28780975
- [Background] Behrendt CA, Riess HC, Schwaneberg T, Larena-Avellaneda A, Kolbel T, Tsilimparis N, Spanos K, Debus ES, Sedrakyan A. Incidence, Predictors, and Outcomes of Colonic Ischaemia in Abdominal Aortic Aneurysm Repair. Eur J Vasc Endovasc Surg. 2018 Oct;56(4):507-513. doi: 10.1016/j.ejvs.2018.06.010. Epub 2018 Jul 20. PMID 30037737
- [Background] Deery SE, O'Donnell TFX, Bodewes TCF, Dalebout BA, Pothof AB, Shean KE, Darling JD, Schermerhorn ML. Early reintervention after open and endovascular abdominal aortic aneurysm repair is associated with high mortality. J Vasc Surg. 2018 Feb;67(2):433-440.e1. doi: 10.1016/j.jvs.2017.06.104. Epub 2017 Sep 21. PMID 28943011
- [Background] Trenner M, Haller B, Storck M, Reutersberg B, Kallmayer MA, Eckstein HH. Trends in Patient Safety of Intact Abdominal Aortic Aneurysm Repair: German Registry Data on 36,594 Procedures. Eur J Vasc Endovasc Surg. 2017 May;53(5):641-647. doi: 10.1016/j.ejvs.2016.12.024. Epub 2017 Jan 19. PMID 28110907
- [Background] Hynes CF, Endicott KM, Iranmanesh S, Amdur RL, Macsata R. Reoperation rates after open and endovascular abdominal aortic aneurysm repairs. J Vasc Surg. 2017 May;65(5):1323-1328. doi: 10.1016/j.jvs.2016.09.053. Epub 2017 Jan 7. PMID 28073669
- [Background] Prinssen M, Verhoeven EL, Buth J, Cuypers PW, van Sambeek MR, Balm R, Buskens E, Grobbee DE, Blankensteijn JD; Dutch Randomized Endovascular Aneurysm Management (DREAM)Trial Group. A randomized trial comparing conventional and endovascular repair of abdominal aortic aneurysms. N Engl J Med. 2004 Oct 14;351(16):1607-18. doi: 10.1056/NEJMoa042002. PMID 15483279
- [Background] Lo RC, Bensley RP, Hamdan AD, Wyers M, Adams JE, Schermerhorn ML; Vascular Study Group of New England. Gender differences in abdominal aortic aneurysm presentation, repair, and mortality in the Vascular Study Group of New England. J Vasc Surg. 2013 May;57(5):1261-8, 1268.e1-5. doi: 10.1016/j.jvs.2012.11.039. Epub 2013 Feb 4. PMID 23384493
- [Background] Wiersema A, Bruijninckx C, Reijnen M, Vos J, Van Delden O, Vahl A, Zeebregts C, Moll F. Perioperative prophylactic antithrombotic strategies in vascular surgery: current practice in the Netherlands. J Cardiovasc Surg (Torino). 2015 Feb;56(1):119-25. Epub 2013 Jan 22. PMID 23337406
- [Background] Wiersema AM, Jongkind V, Bruijninckx CM, Reijnen MM, Vos JA, van Delden OM, Zeebregts CJ, Moll FL; CAPPAStudy Group Consensus on Arterial PeriProcedural Anticoagulation. Prophylactic perioperative anti-thrombotics in open and endovascular abdominal aortic aneurysm (AAA) surgery: a systematic review. Eur J Vasc Endovasc Surg. 2012 Oct;44(4):359-67. doi: 10.1016/j.ejvs.2012.06.008. Epub 2012 Jul 24. PMID 22831869
- [Background] Hirsh J, Raschke R. Heparin and low-molecular-weight heparin: the Seventh ACCP Conference on Antithrombotic and Thrombolytic Therapy. Chest. 2004 Sep;126(3 Suppl):188S-203S. doi: 10.1378/chest.126.3_suppl.188S. PMID 15383472
- [Background] Finley A, Greenberg C. Review article: heparin sensitivity and resistance: management during cardiopulmonary bypass. Anesth Analg. 2013 Jun;116(6):1210-22. doi: 10.1213/ANE.0b013e31827e4e62. Epub 2013 Feb 13. PMID 23408671
- [Background] Arsenault KA, Paikin JS, Hirsh J, Dale B, Whitlock RP, Teoh K, Young E, Ginsberg JS, Weitz JI, Eikelboom JW. Subtle differences in commercial heparins can have serious consequences for cardiopulmonary bypass patients: A randomized controlled trial. J Thorac Cardiovasc Surg. 2012 Oct;144(4):944-950.e3. doi: 10.1016/j.jtcvs.2012.05.065. Epub 2012 Jun 27. PMID 22743176
- [Background] Nath FC, Muller DW, Rosenschein U, Ellis SG, Topol EJ. Heparin monitoring during coronary intervention: activated clotting time versus activated partial thromboplastin time. Can J Cardiol. 1993 Nov;9(9):797-801. PMID 8281479
- [Background] Chew DP, Bhatt DL, Lincoff AM, Moliterno DJ, Brener SJ, Wolski KE, Topol EJ. Defining the optimal activated clotting time during percutaneous coronary intervention: aggregate results from 6 randomized, controlled trials. Circulation. 2001 Feb 20;103(7):961-6. doi: 10.1161/01.cir.103.7.961. PMID 11181470
- [Background] Kasapis C, Gurm HS, Chetcuti SJ, Munir K, Luciano A, Smith D, Aronow HD, Kassab EH, Knox MF, Moscucci M, Share D, Grossman PM. Defining the optimal degree of heparin anticoagulation for peripheral vascular interventions: insight from a large, regional, multicenter registry. Circ Cardiovasc Interv. 2010 Dec;3(6):593-601. doi: 10.1161/CIRCINTERVENTIONS.110.957381. Epub 2010 Nov 9. PMID 21062999
- [Background] Veerhoek D, Groepenhoff F, van der Sluijs MGJM, de Wever JWB, Blankensteijn JD, Vonk ABA, Boer C, Vermeulen CFW. Individual Differences in Heparin Sensitivity and Their Effect on Heparin Anticoagulation During Arterial Vascular Surgery. Eur J Vasc Endovasc Surg. 2017 Oct;54(4):534-541. doi: 10.1016/j.ejvs.2017.07.006. Epub 2017 Aug 9. PMID 28802634
- [Background] Coyne TJ, Wallace MC, Benedict C. Peri-operative anticoagulant effects of heparinization for carotid endarterectomy. Aust N Z J Surg. 1994 Oct;64(10):679-83. doi: 10.1111/j.1445-2197.1994.tb02056.x. PMID 7945064
- [Background] Poisik A, Heyer EJ, Solomon RA, Quest DO, Adams DC, Baldasserini CM, McMahon DJ, Huang J, Kim LJ, Choudhri TF, Connolly ES. Safety and efficacy of fixed-dose heparin in carotid endarterectomy. Neurosurgery. 1999 Sep;45(3):434-41; discussion 441-2. doi: 10.1097/00006123-199909000-00003. PMID 10493364
- [Background] de Sousa AA, Dellaretti MA, Faglioni W Jr, Carvalho GT. Monitoring of activated coagulation time in carotid endarterectomy. Surg Neurol. 2005;64 Suppl 1:S1:6-9. doi: 10.1016/j.surneu.2005.04.016. PMID 15967231
- [Background] Saw J, Bajzer C, Casserly IP, Exaire E, Haery C, Sachar R, Lee D, Abou-Chebl A, Yadav JS. Evaluating the optimal activated clotting time during carotid artery stenting. Am J Cardiol. 2006 Jun 1;97(11):1657-60. doi: 10.1016/j.amjcard.2005.12.062. Epub 2006 Apr 19. PMID 16728233
- [Background] Goldhammer JE, Zimmerman D. Pro: Activated Clotting Time Should Be Monitored During Heparinization For Vascular Surgery. J Cardiothorac Vasc Anesth. 2018 Jun;32(3):1494-1496. doi: 10.1053/j.jvca.2017.04.047. Epub 2017 Apr 26. No abstract available. PMID 28943189
- [Background] Dieplinger B, Egger M, Luft C, Hinterreiter F, Pernerstorfer T, Haltmayer M, Mueller T. Comparison between activated clotting time and anti-activated factor X activity for the monitoring of unfractionated heparin therapy in patients with aortic aneurysm undergoing an endovascular procedure. J Vasc Surg. 2018 Aug;68(2):400-407. doi: 10.1016/j.jvs.2017.11.079. Epub 2018 Mar 20. PMID 29571622
- [Background] Lee JM, Park EY, Kim KM, Won JC, Jung TK, Lee SK. Comparison of activated clotting times measured using the Hemochron Jr. Signature and Medtronic ACT Plus during cardiopulmonary bypass with acute normovolemic haemodilution. J Int Med Res. 2018 Feb;46(2):873-882. doi: 10.1177/0300060517731952. Epub 2017 Oct 4. PMID 28974132
- [Background] Chia S, Van Cott EM, Raffel OC, Jang IK. Comparison of activated clotting times obtained using Hemochron and Medtronic analysers in patients receiving anti-thrombin therapy during cardiac catheterisation. Thromb Haemost. 2009 Mar;101(3):535-40. PMID 19277416
- [Background] Biancari F, Ruggieri VG, Perrotti A, Svenarud P, Dalen M, Onorati F, Faggian G, Santarpino G, Maselli D, Dominici C, Nardella S, Musumeci F, Gherli R, Mariscalco G, Masala N, Rubino AS, Mignosa C, De Feo M, Della Corte A, Bancone C, Chocron S, Gatti G, Gherli T, Kinnunen EM, Juvonen T. European Multicenter Study on Coronary Artery Bypass Grafting (E-CABG registry): Study Protocol for a Prospective Clinical Registry and Proposal of Classification of Postoperative Complications. J Cardiothorac Surg. 2015 Jun 30;10:90. doi: 10.1186/s13019-015-0292-z. PMID 26123033
- [Background] Brascia D, Reichart D, Onorati F, Perrotti A, Ruggieri VG, Bounader K, Verhoye JP, Santarpino G, Fischlein T, Maselli D, Dominici C, Mariscalco G, Gherli R, Rubino AS, De Feo M, Bancone C, Gatti G, Santini F, Dalen M, Saccocci M, Faggian G, Tauriainen T, Kinnunen EM, Nicolini F, Gherli T, Rosato S, Biancari F. Validation of Bleeding Classifications in Coronary Artery Bypass Grafting. Am J Cardiol. 2017 Mar 1;119(5):727-733. doi: 10.1016/j.amjcard.2016.11.027. Epub 2016 Dec 3. PMID 28024656
- [Background] Mazzalai F, Piatto G, Toniato A, Lorenzetti R, Baracchini C, Ballotta E. Using protamine can significantly reduce the incidence of bleeding complications after carotid endarterectomy without increasing the risk of ischemic cerebral events. World J Surg. 2014 May;38(5):1227-32. doi: 10.1007/s00268-013-2347-4. PMID 24276985
- [Background] Yamamoto S, Sakakura K, Taniguchi Y, Yamamoto K, Wada H, Momomura SI, Fujita H. Safety of Reversing Anticoagulation by Protamine Following Elective Transfemoral Percutaneous Coronary Intervention in the Drug-Eluting Stent Era. Int Heart J. 2018 May 30;59(3):482-488. doi: 10.1536/ihj.17-352. Epub 2018 May 9. PMID 29743410
- [Background] Wanhainen A, Verzini F, Van Herzeele I, Allaire E, Bown M, Cohnert T, Dick F, van Herwaarden J, Karkos C, Koelemay M, Kolbel T, Loftus I, Mani K, Melissano G, Powell J, Szeberin Z, Esvs Guidelines Committee, de Borst GJ, Chakfe N, Debus S, Hinchliffe R, Kakkos S, Koncar I, Kolh P, Lindholt JS, de Vega M, Vermassen F, Document Reviewers, Bjorck M, Cheng S, Dalman R, Davidovic L, Donas K, Earnshaw J, Eckstein HH, Golledge J, Haulon S, Mastracci T, Naylor R, Ricco JB, Verhagen H. Editor's Choice - European Society for Vascular Surgery (ESVS) 2019 Clinical Practice Guidelines on the Management of Abdominal Aorto-iliac Artery Aneurysms. Eur J Vasc Endovasc Surg. 2019 Jan;57(1):8-93. doi: 10.1016/j.ejvs.2018.09.020. Epub 2018 Dec 5. No abstract available. PMID 30528142
- [Background] Bellomo R, Ronco C, Kellum JA, Mehta RL, Palevsky P; Acute Dialysis Quality Initiative workgroup. Acute renal failure - definition, outcome measures, animal models, fluid therapy and information technology needs: the Second International Consensus Conference of the Acute Dialysis Quality Initiative (ADQI) Group. Crit Care. 2004 Aug;8(4):R204-12. doi: 10.1186/cc2872. Epub 2004 May 24. PMID 15312219
- [Background] M Versteegh M, M Vermeulen K, M A A Evers S, de Wit GA, Prenger R, A Stolk E. Dutch Tariff for the Five-Level Version of EQ-5D. Value Health. 2016 Jun;19(4):343-52. doi: 10.1016/j.jval.2016.01.003. Epub 2016 Mar 30. PMID 27325326
- [Derived] Wiersema AM, Roosendaal LC, Koelemaij MJW, Tijssen JGP, van Dieren S, Blankensteijn JD, Debus ES, Middeldorp S, Heyligers JMM, Fokma YS, Reijnen MMPJ, Jongkind V. ACTION-1: study protocol for a randomised controlled trial on ACT-guided heparinization during open abdominal aortic aneurysm repair. Trials. 2021 Sep 19;22(1):639. doi: 10.1186/s13063-021-05552-7. PMID 34538275